CLINICAL TRIAL: NCT01992835
Title: Resolution of Allergic Inflammation: Identification and Kinetics of Specific Lipid Mediators During Nasal Allergen Challenge
Brief Title: Resolution of Allergic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 5507
Record Dates: First submitted 2013-10-24; First posted 2013-11-25 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Grass Pollen Allergic Rhinitis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- measurement of mediators in biological fluids (Placebo Comparator)
  Interventions: Other: placebo
- Grass pollen allergen extract (Experimental)
  Interventions: Other: Grass pollen allergen extract

INTERVENTIONS:
Other: Grass pollen allergen extract — Each subject will be challenged with a grass pollen allergen extract and with placebo.
  Arms: Grass pollen allergen extract
Other: placebo
  Arms: measurement of mediators in biological fluids

SUMMARY:
After an allergen challenge, the allergic inflammatory response disappears spontaneously. The initiation of the resolution of the inflammatory response is now recognized as a dynamic process, involving active biochemical programs that enable inflamed tissues to return to homeostasis. Recent data established key roles of different specific lipid mediators in the endogenous counter-regulation of inflammation and activation of resolution. Only little is known about kinetics of these specialized pro-resolving lipid mediators during acute allergic inflammation. Therefore, the primary propose of our study is to characterize the temporal evolution of cellular inflammation and specific lipid mediators after allergen challenge.

ELIGIBILITY:
Eligibility criteria:

Inclusion Criteria

* Allergic rhinitis during the grass pollen season with or without asthma, with at least one of the following symptoms: nasal congestion, itching, rhinorrhea, sneezing
* Grass pollen sensitization determined by a positive skin prick test and / or presence of specific IgEs to a grass pollen allergen extract

Exclusion Criteria:

* Smoker
* Specific immunotherapy with grass allergens or other respiratory allergen for inclusion.
* Current exhibition to another clinically relevant respiratory allergen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Clinical nasal score and measurement of mediators in biological fluids | Measurement of mediators in biological fluids during 72 h after nasal allergen challenge
Clinical nasal score and measurement of mediators in biological fluids. | Measurement and indentification of specific lipid mediators during nasal allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Barnig, Principal Investigator — Pôle de Pathologie Thoracique- Hôpitaux Universitaires Strasbourg
Locations (1):
- Hôpitaux Universitaires, Strasbourg, France

REFERENCES:
- [Result] Qi S, Barnig C, Charles AL, Poirot A, Meyer A, Clere-Jehl R, de Blay F, Geny B. Effect of nasal allergen challenge in allergic rhinitis on mitochondrial function of peripheral blood mononuclear cells. Ann Allergy Asthma Immunol. 2017 Mar;118(3):367-369. doi: 10.1016/j.anai.2016.11.026. Epub 2017 Jan 7. No abstract available. PMID 28073613